CLINICAL TRIAL: NCT00339313
Title: Food Intake and Appetite in the Children of Mothers With Diabetes
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999900005; OH00-DK-N005
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-06-24

CONDITIONS: Diabetes
Keywords: Obesity; Etiology; Macronutrient Selection; Taste Preference; Mixed Meal Test
MeSH Terms: conditions — Diabetes Mellitus; Obesity

SUMMARY:
This protocol is for study of the effect of inhibition of parasympathetic outflow on insulin secretion and glucose metabolism. Insulin secretion will be measured during infusions of escalating doses of atropine. Other clinical parameters of parasympathetic inhibition by atropine will also be assessed.

DETAILED DESCRIPTION:
Children of mothers who had diabetes during pregnancy are at an increased risk of diabetes and obesity in later life, effects partly mediated by the early environment experienced by the offspring of diabetic mothers in utero. In this protocol, we address why intra-uterine exposure to maternal diabetes might lead to later childhood obesity. Previous studies of children of diabetic mothers have not detected any alteration in energy expenditure, either as resting metabolic rate or physical activity. We will now examine whether they are at an increased risk of obesity due to differences in food intake. We will assess composition of the diet, patterns of eating, taste preference and physiological responses to a mixed meal. No previous work in human subjects has addressed these issues.

ELIGIBILITY:
* INCLUSION CRITERIA:

Group 1: Offspring of mothers with diabetes during pregnancy.

Maternal diagnosis of type 2 diabetes (by WHO criteria after a 75g OGTT or on clinical grounds with at least one random plasma glucose greater than 200mg/dl) before or during the index pregnancy.

Group 2: Offspring of mothers with diabetes diagnosed following pregnancy.

Maternal diagnosis of type 2 diabetes (by WHO criteria after a 75g OGTT or on clinical grounds with at least one random plasma glucose greater than 200 mg/dl) after the index pregnancy.

It is important to also ensure that these mothers did not have any major disturbance in glucose tolerance during the index pregnancy and a record of normal glucose tolerance after the index pregnancy; therefore they will only be included if there are also:

Adequate records of glucose testing during the index pregnancy and these records are not in keeping with a diagnosis of gestational diabetes (by either WHO criteria if a 75g oral glucose tolerance test has been carried out).

At least one non-diabetic OGTT after the index pregnancy.

EXCLUSION CRITERIA:

1. History of weight loss for child (greater than 2kg over last 6 months).
2. Presence of other major illnesses which might interfere with appetite or food intake in mother or child.
3. Child not living with mother.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2000-01-12; Study Completion 2011-06-24

CONTACTS AND LOCATIONS:
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Background] Pettitt DJ, Baird HR, Aleck KA, Bennett PH, Knowler WC. Excessive obesity in offspring of Pima Indian women with diabetes during pregnancy. N Engl J Med. 1983 Feb 3;308(5):242-5. doi: 10.1056/NEJM198302033080502. PMID 6848933
- [Background] Silverman BL, Landsberg L, Metzger BE. Fetal hyperinsulinism in offspring of diabetic mothers. Association with the subsequent development of childhood obesity. Ann N Y Acad Sci. 1993 Oct 29;699:36-45. doi: 10.1111/j.1749-6632.1993.tb18835.x. No abstract available. PMID 8267335
- [Background] Pettitt DJ, Aleck KA, Baird HR, Carraher MJ, Bennett PH, Knowler WC. Congenital susceptibility to NIDDM. Role of intrauterine environment. Diabetes. 1988 May;37(5):622-8. doi: 10.2337/diab.37.5.622. PMID 3360218